CLINICAL TRIAL: NCT06440876
Title: Interactive Music And Guided Imagery for Nonpharma Headache Ease
Brief Title: Music and Imagery for Veterans With Migraine Headache
Acronym: IMAGINE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Richard L. Roudebush VA Medical Center (U.S. Federal Agency)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kristin Story, Kristin Maya Story, Richard L. Roudebush VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19092
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music and Imagery (Experimental): MI sessions will be delivered by board-certified music therapists with specialized training in MI and the study treatment protocol. The 8-session protocol has two stages. Stage 1 (sessions 1-4) is focused on learning to use music and imagery for self-regulation. Once the Veteran has demonstrated skill in using music for self-regulation, Stage 2 (sessions 5-8) shifts to identify and deepen their inner resources and how they can use those resources for self-care.
  Interventions: Behavioral: Music and Imagery

INTERVENTIONS:
Behavioral: Music and Imagery — See music and imagery arm description.
  Other Names: MI; Supportive MI

SUMMARY:
The purpose of this study is to determine feasibility and acceptability of telehealth music imagery for migraine (Aim 1) and to explore whether there are clinically meaningful changes in headache frequency and associated patient-centered outcomes (Aim 2).

DETAILED DESCRIPTION:
IMAGINE is a single arm pilot trial. At least 10 and up to 25 Veterans with migraine headache will participate in 8-weekly one-to-one telehealth MI sessions. Sessions will be conducted via a private channel in VA Microsoft Teams, which is a VA approved platform. Each 60-minute MI session is facilitated by a music therapist and consists of 1) a verbal check-in 2) music listening (Veteran patient and therapist choose music together) 3) processing imagery elicited by music, which is done through optional artwork or discussion of the imagery 4) identification of ways to continue to work with music and imagery independently between sessions. Feasibility metrics related to recruitment, retention, engagement, and completion of treatment protocols and assessments will be evaluated. Acceptability will be measured through brief feedback from participant interviews. Qualitative interviews will be conducted to attain Veteran experiences, including perceived benefits, barriers and facilitators. Interview transcripts will be coded and analyzed for emergent themes. Aim 2 outcomes will be explored through changes in headache frequency and associated symptoms from baseline to follow-up immediately following completion of MI sessions. Descriptive statistics will be used to report outcomes. This study is not powered to detect differences in outcomes.

ELIGIBILITY:
Inclusion Criteria:

* A migraine headache ICD-10 diagnosis, and confirmed by the American Migraine Prevalence and Prevention (AMPP) assessment.
* Completion of at least 28 headache diary days
* A confirmed frequency of ≥4 headache days per month
* Confirmed access to a smartphone, computer/tablet
* A primary pain complaint of headache. Patients must be stabilized on their headache medications. Patients must be on their current headache medications for the last 3 months and have no known future changes to those medications for the next 3 months from the start of enrollment.

Exclusion Criteria:

* Non-Veterans
* Veterans without a migraine headache ICD-10 diagnosis
* Veterans without a migraine headache confirmation from AMPP
* Veterans whose primary pain complaint is not headache
* Veterans who do not speak English
* Veterans with a significant cognitive impairment based on EHR ICD10 diagnosis [Mild Cognitive Impairment G31.84; Dementia F03.90; Alzheimer's Dementia G30.9] and confirmed by the Short Portable Mental Status Questionnaire (SPMSQ)19 cognitive screener during the initial baseline assessment. Veterans with a hearing deficit that would impair participation in the MI intervention
* Veterans who have a diagnosis of Traumatic Brain Injury ≤ 1 year before diagnosis of migraine or worsening of migraine as indicated by post-traumatic headache screening tool
* Veterans currently suffering from a disabling psychiatric illness (as noted by clinician); or psychiatric hospitalization in the last 6 months
* Veterans who have active psychotic symptoms, suicidality, or severe depressive symptoms (PHQ score >20) per patient report and/or EHR notes
* Veterans who have had suicidal and/or homicidal ideation in the past 6 months.
* Veterans who decline to or cannot pass the tech screening4b
* Veterans receiving hospice or palliative care
* Veterans who do not have access to smartphone, computer/tablet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility metrics | 2 months
  Percentage of contacted and eligible Veterans consent to study participation, attend intervention sessions, and complete the treatment protocol and scheduled outcome assessments
Acceptability interviews | 6 month
  Veterans will be interviewed after completing study sessions to assess experiences of telehealth MI; aspects of the intervention, especially virtually delivery, that Veterans perceive to be most/least helpful or most/least liked; barriers and facilitators to study participation; how the music interventions compare to other migraine treatments already tried.

SECONDARY OUTCOMES:
Headache Diary | Baseline and 3 months
  Log of headache frequency and characteristics
Music Diary | During active music intervention (months 1-2)
  Log of music listening frequency
Patient Health Questionnaire (PHQ-9) | 3 month
  Depression, self-reported assessment
Migraine Disability Assessment | baseline and 3 month
  5 item self reported assessment for headache-related disability
Veterans RAND 12-item (VR-12) | baseline and 3 month
  12-item, self-report measure of health-related quality life
Generalized Anxiety Disorder Screener (GAD-7) | baseline and 3 month
  7-item, self-report measure of anxiety
Post-Traumatic Stress Disorder Checklist (PCL-5) | baseline and 3 month
  a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD
Headache Pain Catastrophizing Scale (HPCS) | baseline and 3 month
  The HPCS is a 13-item self-report measure of catastrophic thinking related to headache
Headache Management Self-Efficacy Scale (HMSE) | baseline and 3 month
  a 25-item self-report questionnaire related to a person's confidence in their ability to manage their headache symptoms
Patient Global Perception of Change (PGPC) | 3 month
  single item scale measures the participant's perception of improvement since the start of the study

IPD SHARING:
Plan to Share IPD: No